CLINICAL TRIAL: NCT01297322
Title: A Multi-Center, Prospective, Randomized, Controlled, Trial to Evaluate the Safety and Efficacy of the Cardiva VASCADE VCS vs. Manual Compression for the Management of the Femoral Arteriotomy After Percutaneous Endovascular Procedures
Brief Title: RESPECT Trial - (Rapid Extravascular Sealing Via PercutanEous Collagen ImplanT)
Acronym: RESPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiva Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTL 0243
Record Dates: First submitted 2011-02-10; First posted 2011-02-16 (Estimated); Results first posted 2014-10-03 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Surgical Wound
Keywords: vascular closure system; manual compression; femoral arteriotomy; percutaneous endovascular procedures
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual compression (Active Comparator): Using manual compression to reach hemostasis
  Interventions: Other: Manual compression
- VASCADE™ Vascular Closure System (Experimental): The Cardiva VASCADETM Vascular Closure System (VCS) is indicated for the percutaneous closure of common femoral artery access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular catheterization procedures utilizing 6 Fr or 7 Fr procedural sheaths.
  Interventions: Device: Cardiva VASCADE™ Vascular Closure System

INTERVENTIONS:
Other: Manual compression — Standard of Care
  Arms: Manual compression
Device: Cardiva VASCADE™ Vascular Closure System — Investigational Hemostatic Vascular Closure System
  Arms: VASCADE™ Vascular Closure System

SUMMARY:
The objective of this trial is to demonstrate the safety and effectiveness of the Cardiva VASCADE™ Vascular Closure System (VCS) in sealing femoral arterial access sites. Hypothesis: The Cardiva VASCADE™ VCS provides times to hemostasis (TTH) and time to ambulation (TTA) results that are less than manual compression by a clinically meaningful and statistically significant margin. The rate of major access site-related complications with the Cardiva VASCADE™ VCS is non-inferior to the major complication rates of manual compression for sealing femoral arterial access sites.

DETAILED DESCRIPTION:
A prospective, randomized, controlled multi-center clinical trial designed to evaluate the safety and effectiveness of the study device in sealing femoral arterial access sites and providing reduced times to hemostasis and ambulation compared with manual compression at the completion of diagnostic or interventional endovascular procedures performed through 6 Fr or 7 Fr introducer sheaths. Subjects will be randomized in a 2:1 treatment device to control ratio.

ELIGIBILITY:
Pre-Operative Inclusion Criteria:

* Patients undergoing an elective, non-emergent diagnostic or interventional endovascular procedure via the common femoral artery using a 6 or 7 Fr introducer sheath

Pre-Operative Exclusion Criteria:

1. Advanced refusal of blood transfusion, if necessary;
2. Active systemic or a cutaneous infection or inflammation;
3. Pre-existing immunodeficiency disorder and/or chronic use of systemic steroids;
4. Known, significant history of bleeding diathesis, coagulopathy, von Willebrand's disease or current platelet count < 100,000 cells/mm3, baseline INR ≥1.8, or fibrinogen level less than 150 mg/dl (if received a fibrinolytic agent within prior 24 hours);
5. Severe co-existing morbidities having a life expectancy of less than 30 days;
6. Currently involved in any other investigational clinical trial;
7. Ipsilateral femoral arteriotomy within the previous 30 days;
8. Planned endovascular procedure within the next 30 days;
9. Previous ipsilateral femoral artery closure using a permanent implant-based closure device;
10. Previous vascular grafts or surgery at the target vessel access site;
11. History of symptomatic peripheral arterial disease, revascularization or deep vein thrombosis in the ipsilateral limb;
12. Unilateral or bilateral lower extremity amputation(s);
13. Significant anemia with a hemoglobin level less than 10 g/dL or a hematocrit less than 30%;
14. Renal insufficiency (serum creatinine of > 2.5 mg/dl);
15. Females who are pregnant, planning to become pregnant within 3 months of the procedure, or lactating;
16. Extreme morbid obesity (BMI greater than 45 kg/m2) or underweight (BMI less than 20 kg/m2);
17. Unable to routinely walk at least 20 feet without assistance (see protocol);
18. Known allergy/adverse reaction to bovine derivatives, sodium hyaluronate or hyaluronan preparations;
19. Procedures that extend hospitalization (e.g., staged endovascular procedure, CABG);
20. Administration of low molecular weight heparin (LMWH) within 8 hours of the procedure.

Intra-op Exclusion Criteria

1. An introducer sheath with an overall length greater than 11 cm, or not 6 Fr or 7 Fr diameter;
2. Femoral artery diameter less than 6 mm at access site;
3. Difficult insertion of procedural sheath or needle stick problems at the onset of the procedure (e.g., multiple stick attempts, "back wall stick", etc.);
4. Angiographic evidence of more than minimal calcium, atherosclerotic disease, or stent within 1 cm of the puncture site;
5. Overlapping Common Femoral Vein and Femoral Artery at access site;
6. Placement of ipsilateral venous sheath during procedure;
7. Arterial access site located not at common femoral artery (e.g., on or below the bifurcation, above the lower border of the inferior epigastric artery, or above the pelvic brim);
8. More than one access site required;
9. Loss of distal pulses in the ipsilateral extremity during the procedure;
10. Subjects receiving unfractionated heparin with an ACT greater than 300 seconds in the absence of a glycoprotein IIb/IIIa inhibitor or greater than 250 seconds in the presence of a glycoprotein IIb/IIIa inhibitor (may wait to remove introducer sheath until ACT level reaches the target value);
11. Intra-procedural bleeding around sheath, or suspected intraluminal thrombus, hematoma, pseudoaneurysm, or AV fistula;
12. Systemic hypertension (BP greater than 180/110 mmHg) or hypotension (BP less than 90/60 mmHg) prior to randomization;
13. Length of the tissue tract, the distance between the anterior arterial wall and skin, is estimated to be less than 2.5 cm;
14. If the physician deems that a different method should be used to achieve hemostasis of the arterial site or that the subject should not attempt ambulation according to the protocol requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B. Hermiller, Jr., MD, FACC, Principal Investigator — The St. Vincent Heart Center of Indiana, St. Vincent Hospital
Locations (21):
- United States (20):
  - Thomas Hospital, Fairhope, Alabama
  - Christiana Care, Newark, Delaware
  - Holmes Regional Medical Center, Melbourne, Florida
  - St. John's Prairie Heart, Springfield, Illinois
  - St. Vincent's Heart Center of Indiana, Indianapolis, Indiana
  - King's Daughters Medical Center, Ashland, Kentucky
  - Terrebonne General Medical Center, Houma, Louisiana
  - Lafayette General Medical Center, Lafayette, Louisiana
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Tufts University, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Cooper Health System, Camden, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - New York-Presbyterian Hospital, New York, New York
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Heart Hospital of Austin, Austin, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - CAMC Health Education and Research Institute, Inc., Charleston, West Virginia
- St. Vincent's Hospital Melbourne, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Lehmann KG, Heath-Lange SJ, Ferris ST. Randomized comparison of hemostasis techniques after invasive cardiovascular procedures. Am Heart J. 1999 Dec;138(6 Pt 1):1118-25. doi: 10.1016/s0002-8703(99)70078-5. PMID 10577443
- [Background] Simon A, Bumgarner B, Clark K, Israel S. Manual versus mechanical compression for femoral artery hemostasis after cardiac catheterization. Am J Crit Care. 1998 Jul;7(4):308-13. PMID 9656045
- [Background] Kussmaul WG 3rd, Buchbinder M, Whitlow PL, Aker UT, Heuser RR, King SB, Kent KM, Leon MB, Kolansky DM, Sandza JG Jr. Rapid arterial hemostasis and decreased access site complications after cardiac catheterization and angioplasty: results of a randomized trial of a novel hemostatic device. J Am Coll Cardiol. 1995 Jun;25(7):1685-92. doi: 10.1016/0735-1097(95)00101-9. PMID 7759724
- [Background] Castaneda F, Swischuk JL, Smouse HB, Brady T. Gelatin sponge closure device versus manual compression after peripheral arterial catheterization procedures. J Vasc Interv Radiol. 2003 Dec;14(12):1517-23. doi: 10.1097/01.rvi.0000099530.29957.dd. PMID 14654485
- [Background] Hoffer EK, Bloch RD. Percutaneous arterial closure devices. J Vasc Interv Radiol. 2003 Jul;14(7):865-85. doi: 10.1097/01.rvi.0000071086.76348.8e. PMID 12847195
- [Background] Gerckens U, Cattelaens N, Lampe EG, Grube E. Management of arterial puncture site after catheterization procedures: evaluating a suture-mediated closure device. Am J Cardiol. 1999 Jun 15;83(12):1658-63. doi: 10.1016/s0002-9149(99)00174-5. PMID 10392872
- [Background] Kinnaird TD, Stabile E, Mintz GS, Lee CW, Canos DA, Gevorkian N, Pinnow EE, Kent KM, Pichard AD, Satler LF, Weissman NJ, Lindsay J, Fuchs S. Incidence, predictors, and prognostic implications of bleeding and blood transfusion following percutaneous coronary interventions. Am J Cardiol. 2003 Oct 15;92(8):930-5. doi: 10.1016/s0002-9149(03)00972-x. PMID 14556868
- [Background] Newcombe RG. Interval estimation for the difference between independent proportions: comparison of eleven methods. Stat Med. 1998 Apr 30;17(8):873-90. doi: 10.1002/(sici)1097-0258(19980430)17:83.0.co;2-i. PMID 9595617

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Manual Compression | VASCADE™ Vascular Closure System
Started | 142 | 278
Completed | 141 | 274
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Compression | VASCADE™ Vascular Closure System | Total
Number analyzed (Participants) | 142 | 275 | 417
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (10.4) | 61.8 (11.2) | 62 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 79 | 120
  Male | 101 | 196 | 297
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 6 | 18 | 24
  White | 130 | 249 | 379
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Hemostasis (TTH)
Description: Primary effectiveness endpoint - elapsed time between device (VASCADE) or sheath (manual compression) removal and first observed and confirmed arterial hemostasis.
Time Frame: Up to 1 hour
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Manual Compression | VASCADE™ Vascular Closure System
Number analyzed (Participants) | 142 | 275
minutes | 21.4 (12.4) | 4.8 (5.4)

2. Primary Outcome: Rate of Combined Access Site-related Major Complications
Description: Primary safety endpoint
  * Access site-related bleeding requiring transfusion;
  * Vascular injury requiring repair (via surgery, ultrasound guided compression, transcatheter embolization or stent graft);
  * New ipsilateral lower extremity ischemia causing a threat to the viability of the limb and requiring surgical or additional percutaneous intervention. This compromised blood flow is documented by subject symptoms, physical exam and/or a decreased or absent blood flow on lower extremity angiogram.;
  * Access site-related infection requiring intravenous antibiotics and/or extended hospitalization;
  * New onset access site-related neuropathy in the ipsilateral lower extremity requiring surgical repair;
  * Permanent access site-related nerve injury. (> 30 days)
Time Frame: 30 days +/- 7 days
Measure: Number; unit: participants
Arm/Group | Manual Compression | VASCADE™ Vascular Closure System
Number analyzed (Participants) | 142 | 275
participants | 0 | 0

3. Secondary Outcome: Time to Ambulation (TTA)
Description: Secondary effectiveness endpoint - elapsed time between device (VASCADE) or sheath (manual compression) removal and when subject stands and walks 20 feet without evidence of arterial re-bleeding
Time Frame: Up to 1 day
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Manual Compression | VASCADE™ Vascular Closure System
Number analyzed (Participants) | 142 | 275
hours | 5.8 (3.1) | 3.8 (5.1)

4. Secondary Outcome: Time to Discharge Eligibility (TTDE)
Description: Secondary effectiveness endpoint - elapsed time between device (VASCADE) or sheath (manual compression) removal and when subject is medically able to be discharged based solely on the assessment of the access site, as determined by the medical team
Time Frame: Up to 2 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Manual Compression | VASCADE™ Vascular Closure System
Number analyzed (Participants) | 142 | 274
hours | 6.5 (3.3) | 4.8 (6.4)

5. Secondary Outcome: Time to Hospital Discharge (TTHD)
Description: Secondary effectiveness endpoint - elapsed time between device (VASCADE) or sheath (manual compression) removal and when subject is actually discharged from the hospital
Time Frame: Up to 2 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Manual Compression | VASCADE™ Vascular Closure System
Number analyzed (Participants) | 142 | 275
hours | 13.7 (9.8) | 18.3 (34.5)

6. Secondary Outcome: Device Success
Description: Secondary effectiveness endpoint - ability to deploy the delivery system, deliver the collagen, and achieve hemostasis with VASCADE alone or with adjunctive compression
Time Frame: Up to 1 day
Measure: Number; unit: participants
Arm/Group | VASCADE™ Vascular Closure System
Number analyzed (Participants) | 275
participants | 263

7. Secondary Outcome: Procedure Success
Description: Secondary effectiveness endpoint - attainment of final hemostasis using any method and freedom from major vascular complications through 30 days
Time Frame: 30 days +/- 7 days
Measure: Number; unit: participants
Arm/Group | Manual Compression | VASCADE™ Vascular Closure System
Number analyzed (Participants) | 142 | 275
participants | 142 | 275

8. Secondary Outcome: Rate of Combined Minor Access Site Complications
Description: Secondary safety endpoint
  * Access site-related bleeding requiring greater than 30 minutes to achieve hemostasis;
  * Access site-related hematoma > 6 cm;
  * Late access site-related bleeding (following hospital discharge);
  * Ipsilateral lower extremity arterial emboli;
  * Ipsilateral deep vein thrombosis;
  * Access site-related vessel laceration;
  * Access site wound dehiscence;
  * Localized access site infection treated with intramuscular or oral antibiotics;
  * Arteriovenous fistula not requiring treatment;
  * Pseudoaneurysm requiring thrombin injection or fibrin adhesive injection;
  * Pseudoaneurysm not requiring treatment;
  * New onset access site-related neuropathy in the ipsilateral lower extremity not requiring surgical repair;
  * Ipsilateral pedal pulse diminished by two grades or transiently lost.
Time Frame: 30 days +/- 7 days
Measure: Number; unit: participants
Arm/Group | Manual Compression | VASCADE™ Vascular Closure System
Number analyzed (Participants) | 142 | 275
participants | 10 | 3

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Manual Compression | VASCADE™ Vascular Closure System
Serious Adverse Events (participants affected / at risk) | 0/142 | 0/275
Other Adverse Events (participants affected / at risk) | 28/142 | 56/275
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Manual Compression (N=142) | VASCADE™ Vascular Closure System (N=275)
Arterial Thrombosis - peripheral/ non-access site-related (Vascular disorders) | 0 (0) | 1 (1) — Arterial Thrombosis - peripheral/ non-access site-related
Embolization - peripheral non-access site-related (Vascular disorders) | 0 (0) | 1 (1) — Embolization - peripheral non-access site-related
Severe Hypotension Requiring Treatment (Cardiac disorders) | 0 (0) | 3 (3) — Severe Hypotension Requiring Treatment
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Anemia
Renal Insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0) — Renal Insufficiency
Access site re-bleeding after initial hemostasis confirmed for 5 minutes (Blood and lymphatic system disorders) | 4 (4) | 7 (7) — Access site re-bleeding after initial hemostasis confirmed for 5 minutes
Altered mental status (Psychiatric disorders) | 0 (0) | 4 (4) — Altered mental status
Access site-related tissue tract oozing - prolonged (Surgical and medical procedures) | 0 (0) | 1 (1) — Access site-related tissue tract oozing - prolonged
Angina (Cardiac disorders) | 1 (1) | 3 (3) — Angina
Atrial fibrillation (Cardiac disorders) | 0 (0) | 4 (4) — Atrial fibrillation
Cardiac disorders/symptoms (Cardiac disorders) | 0 (0) | 3 (3) — Cardiac disorders/symptoms
Dermatologic disorders / symptoms (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) — Dermatologic disorders / symptoms
Discomfort - access site (Surgical and medical procedures) | 0 (0) | 6 (6) — Discomfort - access site
Discomfort - nonaccess site (General disorders) | 1 (1) | 0 (0) — Discomfort - nonaccess site
Dizziness (General disorders) | 0 (0) | 1 (1) — Dizziness
ENT disorders/symptoms (Ear and labyrinth disorders) | 0 (0) | 1 (1) — ENT disorders/symptoms
Ecchymosis - access site (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Ecchymosis - access site
Ecchymosis - nonaccess site (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Ecchymosis - nonaccess site
Erythema - access site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Erythema - access site
Fall (General disorders) | 0 (0) | 1 (1) — Fall
GI disorders/symptoms (Gastrointestinal disorders) | 4 (4) | 5 (5) — GI disorders/symptoms
GU disorders/symptoms (Renal and urinary disorders) | 0 (0) | 2 (2) — GU disorders/symptoms
General disorder/respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — General disorder/respiratory
General disorders/symptoms (General disorders) | 2 (2) | 4 (4) — General disorders/symptoms
Headache (General disorders) | 4 (4) | 1 (1) — Headache
Hematoma - access site (Blood and lymphatic system disorders) | 2 (2) | 6 (6) — Hematoma - access site
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) — Hematuria
Hypertension (Cardiac disorders) | 1 (1) | 1 (1) — Hypertension
Hypervolemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Hypervolemia
Hypotension (Cardiac disorders) | 1 (1) | 3 (3) — Hypotension
Infection - access site (Infections and infestations) | 0 (0) | 1 (1) — Infection - access site
Neuro - other (Nervous system disorders) | 1 (1) | 2 (2) — Neuro - other
Neurological deficit - TIA (Nervous system disorders) | 0 (0) | 1 (1) — Neurological deficit - TIA
Ortho disorders/symptoms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Ortho disorders/symptoms
Pain - access site (General disorders) | 3 (3) | 2 (2) — Pain - access site
Pain - nonaccess site (General disorders) | 2 (2) | 6 (6) — Pain - nonaccess site
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) — Rash
Renal failure/insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1) — Renal failure/insufficiency
Respiratory disorders/symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) — Respiratory disorders/symptoms
Retroperitoneal bleeding (hematoma/hemorrhage) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Retroperitoneal bleeding (hematoma/hemorrhage)
Swelling - nonaccess site (General disorders) | 0 (0) | 1 (1) — Swelling - nonaccess site
Vascular repair - non-device related (Vascular disorders) | 0 (0) | 1 (1) — Vascular repair - non-device related
Vasovagal episode (Nervous system disorders) | 2 (2) | 1 (1) — Vasovagal episode
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) — Ventricular arrhythmia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-07-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT01297322/Prot_SAP_000.pdf